CLINICAL TRIAL: NCT00936793
Title: Drug Interaction Study Between Inhaled Beclomethasone and Protease Inhibitors in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Scott R. Penzak, Pharm.D./NIH Clinical Center, National Institutes of Health
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 090186; 09-CC-0186
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-02-09

CONDITIONS: HIV; Asthma
Keywords: Drug Interaction; Asthma; HIV; Beclomethasone; Protease Inhibitors; HV; Healthy Volunteer; HIV Infections
MeSH Terms: conditions — Asthma; HIV Infections | interventions — Darunavir; Ritonavir

INTERVENTIONS:
Drug: Darunavir
Drug: Ritonavir
Drug: Beclomethasone Dipropionate HFA

SUMMARY:
Patients with human immunodeficiency virus (HIV) and respiratory disease commonly require protease inhibitors (PIs) and orally inhaled corticosteroids. Inhaled corticosteroids alone do not generally cause systemic adverse effects because of low systemic bioavailability, but the combination of inhaled fluticasone and various PIs has led to increased systemic fluticasone levels and multiple cases of secondary adrenal insufficiency. A study in healthy volunteers showed > 350-fold increase in fluticasone area under the curve when ritonavir (RTV) 100mg twice daily was coadministered with intranasal fluticasone compared to intranasal fluticasone alone. The mechanism of this drug interaction is presumably secondary to PI inhibition of cytochrome P450 3A4, the enzyme responsible for fluticasone metabolism. As a result, inhaled fluticasone is not recommended in combination with most PIs unless the benefit outweighs the risk. One possible alternative to fluticasone is inhaled beclomethasone, which has not been studied in combination with PIs. Although beclomethasone also undergoes metabolism via CYP3A4 in vitro to its more active metabolite, beclomethasone-17-monopropionate, it appears to be largely hydrolyzed by esterases in vivo. Furthermore, the pharmacokinetic properties of beclomethasone-17-monopropionate, such as relatively short half-life, low maximum plasma concentration, and low volume of distribution, suggest that systemic accumulation leading to significant adverse effects is unlikely even in the presence of a CYP3A4 inhibitor such as a PI.

In this open-label study, 46 subjects will receive inhaled beclomethasone for 6 weeks from Days 1 to 42. Subjects will be randomized into 1 of 3 groups, such that from Days 15 to 42, 18 subjects will add no additional study drugs, 14 subjects will add RTV 100mg twice daily, and 14 subjects will add DRV/r 600/100mg twice daily. Pharmacokinetic sampling for beclomethasone and beclomethasone-17-monopropionate levels will occur on Days 14 and 28. Pre-cosyntropin cortisol levels and a low-dose adrenocorticotropic hormone (ACTH) stimulation test will be performed on all subjects on Days 1, 14, 28, and 42. Data from this investigation will determine whether RTV and/or DRV/r, potent CYP 3A4 inhibitors, alter the pharmacokinetics of beclomethasone and its active metabolite, beclomethasone-17-monopropionate (primary objective), and whether or not a possible increase in systemic bioavailability of beclomethasone and beclomethasone-17-monopropionate alters pre-cosyntropin cortisol levels and responses to ACTH stimulation test over a 4-week period (secondary objective). Results from this investigation will provide pharmacokinetic and pharmacodynamic data to assist clinicians in determining whether inhaled beclomethasone is an appropriate option in HIV-infected patients requiring concomitant therapy with an inhaled corticosteroid and PIs.

DETAILED DESCRIPTION:
Patients with human immunodeficiency virus (HIV) and respiratory disease commonly require protease inhibitors (PIs) and orally inhaled corticosteroids. Inhaled corticosteroids alone do not generally cause systemic adverse effects because of low systemic bioavailability, but the combination of inhaled fluticasone and various PIs has led to increased systemic fluticasone levels and multiple cases of secondary adrenal insufficiency. A study in healthy volunteers showed > 350-fold increase in fluticasone area under the curve when ritonavir (RTV) 100mg twice daily was coadministered with intranasal fluticasone compared to intranasal fluticasone alone. The mechanism of this drug interaction is presumably secondary to PI inhibition of cytochrome P450 3A4, the enzyme responsible for fluticasone metabolism. As a result, inhaled fluticasone is not recommended in combination with most PIs unless the benefit outweighs the risk. One possible alternative to fluticasone is inhaled beclomethasone, which has not been studied in combination with PIs. Although beclomethasone also undergoes metabolism via CYP3A4 in vitro to its more active metabolite, beclomethasone-17-monopropionate, it appears to be largely hydrolyzed by esterases in vivo. Furthermore, the pharmacokinetic properties of beclomethasone-17-monopropionate, such as relatively short half-life, low maximum plasma concentration, and low volume of distribution, suggest that systemic accumulation leading to significant adverse effects is unlikely even in the presence of a CYP3A4 inhibitor such as a PI.

In this open-label study, 30 subjects will receive inhaled beclomethasone for 6 weeks from Days 1 to 42. Subjects will be randomized into 1 of 3 groups, such that from Days 15 to 42, 10 subjects will add no additional study drugs, 10 subjects will add RTV 100mg twice daily, and 10 subjects will add DRV/r 600/100mg twice daily. Pharmacokinetic sampling for beclomethasone and beclomethasone-17-monopropionate levels will occur on Days 14 and 28. Pre-cosyntropin cortisol levels and a low-dose adrenocorticotropic hormone (ACTH) stimulation test will be performed on all subjects on Days 1, 14, 28, and 42. Data from this investigation will determine whether RTV and/or DRV/r, potent CYP 3A4 inhibitors, alter the pharmacokinetics of beclomethasone and its active metabolite, beclomethasone-17-monopropionate (primary objective), and whether or not a possible increase in systemic bioavailability of beclomethasone and beclomethasone-17-monopropionate alters pre-cosyntropin cortisol levels and responses to ACTH stimulation test over a 4-week period (secondary objective). Results from this investigation will provide pharmacokinetic and pharmacodynamic data to assist clinicians in determining whether inhaled beclomethasone is an appropriate option in HIV-infected patients requiring concomitant therapy with an inhaled corticosteroid and PIs.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Males and females between the ages of 18 and 60 years
  2. Healthy by medical history and physical examination
  3. Laboratory values within established guidelines for participation in clinical studies: aspartate transaminase (AST) less than or equal to 2 times the ULN; serum creatinine less than or equal to the ULN; hemoglobin greater than or equal to 11 g/dL (for both males and females)
  4. Negative serum or urine pregnancy test for females of child-bearing potential
  5. Females of child-bearing potential who are able and willing to practice abstinence or use non-hormonal effective methods of birth control during the study, such as condoms or diaphragms

EXCLUSION CRITERIA:

1. Concomitant routine therapy with any prescription, over-the-counter, herbal, or holistic medications, including hormonal contraceptives by any route, any corticosteroid by any route, any inhaled medications, and any investigational drugs, for 30 days prior to study participation. An exception to this requirement is the use of topical medications that are not significantly absorbed systemically, e.g. topical minoxidil.

   * Concomitant therapy (chronic or intermittent) with any prescription, over-the-counter, or herbal drugs will not be allowed during the study duration
   * Intermittent use of acetaminophen, non-steroidal anti-inflammatory medications (i.e., ibuprofen), and loperamide will be allowed to be taken according to each manufacturer's recommendations during the study, but should not be taken on the days of pharmacokinetic blood sampling
   * A daily multivitamin with minerals will be allowed during the study
   * Use of topical medications that are not significantly absorbed systemically wil be allowed if approved by the Principal Investigator.
2. Inability to obtain venous access for blood sample collection
3. The presence or history of any of the following:

   * adrenal disease (e.g., Addison's disease, Cushing's syndrome, etc.),
   * diabetes mellitus (clinical diagnosis based on current guidelines),
   * HIV infection,
   * pulmonary disease (e.g., asthma, chronic obstructive pulmonary disease, etc.),
   * cardiac disease (e.g., hypertension [systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg], heart failure, arrhythmia, etc.),
   * renal disease (chronic or acute renal failure or insufficiency),
   * hepatitis (as assessed by patient interview) or hepatic impairment,
   * pancreatitis,
   * bleeding disorders (e.g., hemophilia),
   * internal bleeding (such as gastrointestinal or intracranial),
   * peptic ulcer disease requiring maintenance pharmacologic therapy,
   * osteoporosis,
   * osteonecrosis,
   * atopy or atopic dermatitis,
   * hormone-sensitive cancers or conditions,
   * malignancy,
   * organ transplant,
   * seizure disorders,
   * schizophrenia or other psychiatric illnesses that may interfere with the subject's ability to participate in the study, or
   * any other condition that may interfere with the interpretation of the study results or not be in the best interest of the subject in the opinion of the investigators.
4. Baseline cortisol level less than 5 mcg/dL
5. Positive serum or urine pregnancy test or breastfeeding female
6. The presence of persistent diarrhea or malabsorption that would interfere with the subject's ability to absorb drugs
7. Drug or alcohol abuse that may impair safety or adherence
8. History of intolerance or allergic reaction to darunavir, ritonavir, beclomethasone, cosyntropin, or any inhaled medication
9. Fasting total cholesterol greater than 240 mg/dL or fasting triglycerides greater than 400 mg/dL
10. Fasting glucose greater than100 mg/dL
11. Use of nicotine-containing tobacco products, including cigarettes and chewing tobacco

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2009-07-06; Primary Completion 2011-06-10 (Actual); Study Completion 2011-06-10 (Actual)

PRIMARY OUTCOMES:
Influence of Darunavir/Ritonavir and Ritonavir alone on the pharmacokinetics of inhaled Beclomethasone.

SECONDARY OUTCOMES:
Alterations in renal function in healthy subjects receiving inhaled Beclomethasone alone and with HIV protease inhibitors

CONTACTS AND LOCATIONS:
Overall Officials: Susan F Leitman, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Foisy MM, Yakiwchuk EM, Chiu I, Singh AE. Adrenal suppression and Cushing's syndrome secondary to an interaction between ritonavir and fluticasone: a review of the literature. HIV Med. 2008 Jul;9(6):389-96. doi: 10.1111/j.1468-1293.2008.00579.x. Epub 2008 May 4. PMID 18459946
- [Background] Clevenbergh P, Corcostegui M, Gerard D, Hieronimus S, Mondain V, Chichmanian RM, Sadoul JL, Dellamonica P. Iatrogenic Cushing's syndrome in an HIV-infected patient treated with inhaled corticosteroids (fluticasone propionate) and low dose ritonavir enhanced PI containing regimen. J Infect. 2002 Apr;44(3):194-5. doi: 10.1053/jinf.2001.0928. PMID 12099750
- [Background] Rouanet I, Peyriere H, Mauboussin JM, Vincent D. Cushing's syndrome in a patient treated by ritonavir/lopinavir and inhaled fluticasone. HIV Med. 2003 Apr;4(2):149-50. doi: 10.1046/j.1468-1293.2003.00149.x. No abstract available. PMID 12702137